CLINICAL TRIAL: NCT06315504
Title: Circulating Factors in Nephrotic Syndrome - A Prospective Observational Cohort Study
Brief Title: Circulating Factors in Nephrotic Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Iain Bressendorff (Other)
Responsible Party: Sponsor-Investigator, Iain Bressendorff, MD PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: Nephrotic Syndrome Cohort
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Nephrotic Syndrome; Membranous Nephropathy; Minimal Change Disease; Primary Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulonephritis, Membranous; Nephrosis, Lipoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood and kidney tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with de novo nephrotic syndrome
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
A prospective observational study to investigate the treatment-associated changes of circulating factors associated with glomerular diseases among patients with de novo nephrotic syndrome admitted to hospital for a kidney biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Plasma albumin < 36 g/L
* Urine protein >3.5 g/day or urine protein/creatinine-ratio (UPCR) > 3.5 or urine albumin/creatinine-ratio (UACR) >2200 mg/g
* Planned kidney biopsy
* Able to give written informed consent

Exclusion Criteria:

* Kidney transplant recipient
* Previously undergone a kidney biopsy
* Unable to understand written information in Danish

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: De novo nephrotic syndrome admitted to hospital for a clinically indicated kidney biopsy.
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2034-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
levels of anti-nephrin in blood by ELISA | up to 12 months
  temporal association of anti-nephrin with clinical remission of nephrotic syndrome

SECONDARY OUTCOMES:
changes in auto-antibodies in blood associated with membranous nephropathy | up to 24 months
  temporal association of auto-antibodies with clinical remission of nephrotic syndrome

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request to the primary investigator.